CLINICAL TRIAL: NCT04435782
Title: A Prospective, Multicenter, Single-Arm, Open-Label, Phase 4 Study of the Effects of Selexipag on Right Ventricular Remodeling in Pulmonary Arterial Hypertension Assessed by Cardiac Magnetic Resonance Imaging
Brief Title: A Study of Selexipag Assessing Right Ventricular Remodeling in Pulmonary Arterial Hypertension by Cardiac Magnetic Resonance Imaging
Acronym: RESTORE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The Sponsor decided to prematurely terminate the study due to the lower-than-expected recruitment rate.
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108753; 67896049PAH4005 (Other: Actelion); 2019-004783-22 (EudraCT Number)
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Right ventricle; Reverse remodeling; Magnetic resonance Imaging
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — selexipag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-67896049 (Experimental): Participants will receive JNJ-67896049 tablets at a starting dose of 200 mcg on Day 1. Dose will be up-titrated from Day 1 to the end of Week 12 (Day 84) to determine individual maintenance dose (IMD). Then, participants will receive JNJ-67896049 tablets at their IMD from Week 13 to Week 52.
  Interventions: Drug: JNJ-67896049

INTERVENTIONS:
Drug: JNJ-67896049 — Participants will receive tablets at a starting dose of 200 mcg on Day 1. Dose will be up-titrated from Day 1 to the end of Week 12 (Day 84) to determine individual maintenance dose (IMD). Then, participants will receive JNJ-67896049 tablets at their IMD from Week 13 to Week 52.
  Other Names: Selexipag

SUMMARY:
The purpose of the study is to assess the effects of selexipag on right ventricular (RV) function in participants with Pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* World health organization functional class (WHO FC) II or III. Enrollment will be stratified by WHO FC II or III. Proportion of participants with WHO FC II and WHO FC III are expected to be approximately 40 percent (%) and 60%, respectively
* Pulmonary arterial hypertension (PAH) etiology belonging to one of the following groups according to 6th world symposium of pulmonary hypertension (WSPH) classification: a) Idiopathic PAH, b) Heritable PAH, c) Drugs or toxins induced d) PAH associated with connective tissue disease, e) PAH associated with congenital heart disease, with simple systemic-to-pulmonary shunt at least 1 year after surgical repair
* Patients already receiving PAH-specific oral mono or dual therapy (that is, phosphodiesterase type 5 inhibitors [PDE-5i] or soluble guanylate cyclase stimulators [sGCs] and/or endothelin receptor antagonist [ERA]) or patients who are not candidates for these therapies
* N-terminal-pro-hormone brain natriuretic peptide (NT-proBNP) greater than or equal to (>=) 300 nanograms per liter (ng/L) (greater than or equal to [>=] 300 picograms per milliliter [pg/mL]; >=35.5 picomoles per liter [pmol/L]) at screening
* Women of childbearing potential must meet the following criteria: a) Have a negative serum pregnancy test during screening and a negative urine pregnancy test on Day 1, b) Agree to use acceptable methods of contraception from Day 1 to at least 30 days after study intervention discontinuation, c) If only using hormonal contraception, have used it for at least 1 month (30 days) before Day 1, and d) Agree to perform monthly pregnancy tests to at least 30 days after study intervention discontinuation
* 6-minute walking distance (6MWD) >=150 meter (m) during screening period

Exclusion Criteria:

* Prior use of Prostacyclin (IP)-receptor agonist, prostacyclin, or prostacyclin analog. Use of such treatments for vasoreactivity testing is not exclusionary; intermittent use of such treatments for digital ulcers or Raynaud's phenomenon is not exclusionary if stopped > 6 months (180 days) prior to Day 1
* Treatment with strong inhibitors of CYP2C8 (example, gemfibrozil) within 4 weeks (28 days) prior to Day 1
* Treatment with another investigational drug planned or taken within 12 weeks (84 days) prior to Day 1
* Severe coronary heart disease or unstable angina
* Cerebrovascular events (example, transient ischemic attack, stroke) within 3 months (90 days) prior to Day 1

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (35):
- United States (3):
  - University Of California San Diego, La Jolla, California
  - AnMed Health, Anderson, South Carolina
  - UT Southwestern, Dallas, Texas
- Argentina (3):
  - Hospital Italiano de Buenos Aires, Caba
  - Sanatorio Ramon Cereijo, Caba
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
- Brazil (4):
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - SPDM - Associacao Paulista para o Desenvolvimento da Medicina - Hospital Sao Paulo, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- CHU Grenoble, La Tronche, France
- Germany (3):
  - DRK Kliniken Westend, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
- Hong Kong (2):
  - Grantham Hospital, Hong Kong
  - Queen Mary Hospital University of Hong Kong, Hong Kong
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center Beilinson Campus, Petah Tikva
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Netherlands (2):
  - VUMC Amsterdam, Amsterdam
  - Radboud Umcn, Nijmegen
- Russia (2):
  - National Medical Research Center of Cardiology of MoH of Russian Federation, Moscow
  - Federal State Budgetary Institution, Saint Petersburg
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
- Singapore (2):
  - National Heart Centre (NHC) Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (5):
  - Chungnam National University Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates
- United Kingdom (3):
  - Golden Jubilee National Hospital, Glasgow
  - Royal Free Hospital, Hampstead
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Selexipag: Participants with pulmonary arterial hypertension (PAH) received a 200 microgram (mcg) selexipag tablet orally on the evening of Day 1, followed by twice-daily dosing starting from Day 2. The dose of selexipag was increased by 200 mcg each week to allow each participant to reach their individual maximum dose (iMD), up to 1600 mcg twice daily, by the end of Week 12. From Week 13 onwards, participants received their iMD of 1600 mcg selexipag tablets orally twice daily until Week 52. Participants were then followed for safety up to 30 days after the last dose of selexipag.
Period: Overall Study
Arm/Group | Selexipag
Started | 9
Completed | 5
Not Completed | 4
Not completed — Study terminated by sponsor | 4

BASELINE CHARACTERISTICS:
Arm/Group | Selexipag
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (13.28) [lower limit 13.28]
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 0
  Children (2-11 years) | 0
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 9
  From 65-84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Right Ventricular Stroke Volume (RVSV) Assessed by Pulmonary Artery Flow Magnetic Resonance Imaging (MRI)
Description: Change from baseline to Week 26 in RVSV assessed by pulmonary artery flow MRI was reported.
Time Frame: Baseline, Week 26
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and "n" (Number Analyzed) signifies participants evaluable for specified rows. As pre-specified in the statistical analysis plan (SAP), participant wise data was collected and reported due to very limited number of participants enrolled.
Measure: Number; unit: Milliliter (mL)
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Milliliter (mL)
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 38.35
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | -1.53
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 16.53
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 11
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 27.2
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 14.07

2. Secondary Outcome: Change From Baseline to Week 26 in Right Ventricular End-Diastolic Volume (RVEDV) Assessed by MRI
Description: Change from baseline to Week 26 in RVEDV assessed by MRI was reported.
Time Frame: Baseline, Week 26
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure and "n" (Number Analyzed) signifies participants evaluable for specified rows. As pre-specified in the SAP, participant wise data was collected and reported due to very limited number of participants enrolled.
Measure: Number; unit: Milliliter
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Milliliter
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 40.57
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | -8.89
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 23.58
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 6.79
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 3.71
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 7.82

3. Secondary Outcome: Change From Baseline to Week 26 in Right Ventricular End-Systolic Volume (RVESV) Assessed by MRI
Description: Change from baseline to Week 26 in RVESV assessed by MRI was reported.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Milliliter
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Milliliter
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 2.23
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | -7.36
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 7.05
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | -4.22
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | -23.5
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | -6.25

4. Secondary Outcome: Change From Baseline to Week 26 in Right Ventricular Ejection Fraction (RVEF) Assessed by MRI
Description: Change from baseline to Week 26 in RVEF assessed by MRI was reported. RVEF was the fraction of the end-diastolic volume (EDV) that is ejected out of right ventricle with each contraction. EDV is the volume of blood within a ventricle immediately before a contraction.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Percentage of EDV
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Percentage of EDV
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 9.65
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0.42
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 6.96
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 5.01
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 19.12
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 7.62

5. Secondary Outcome: Change From Baseline to Week 26 in Right Ventricular (RV) Mass Index Assessed by MRI
Description: Change from baseline to Week 26 in RV mass index assessed by MRI was reported.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Grams per meter square (g/m^2)
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Grams per meter square (g/m^2)
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | -11.03
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 2.72
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | -12.69
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 0.09
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | -16.56
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | -2.41

6. Secondary Outcome: Change From Baseline to Week 26 in Right Ventricular Global Longitudinal Strain (RVGLS) Assessed by MRI
Description: Change in RVGLS was a measure of longitudinal percent change in length of endocardium at Week 26 from baseline length assessed by MRI.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Percent change in length of endocardium
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Percent change in length of endocardium
  Participant 1: RVGLS Endocardium: number analyzed (Participants) | 1
  Participant 1: RVGLS Endocardium | -4.26
  Participant 2: RVGLS Endocardium: number analyzed (Participants) | 1
  Participant 2: RVGLS Endocardium | -5.31
  Participant 3: RVGLS Endocardium: number analyzed (Participants) | 1
  Participant 3: RVGLS Endocardium | -12.8
  Participant 4: RVGLS Endocardium: number analyzed (Participants) | 1
  Participant 4: RVGLS Endocardium | -5.61
  Participant 5: RVGLS Endocardium: number analyzed (Participants) | 1
  Participant 5: RVGLS Endocardium | -14.45
  Participant 6: RVGLS Endocardium: number analyzed (Participants) | 1
  Participant 6: RVGLS Endocardium | -1.74

7. Secondary Outcome: Number of Participants With Change From Baseline to Week 26 in World Health Organization (WHO) Functional Class
Description: WHO functional classification for PAH ranged from Class I (no limitation in physical activity, ordinary physical activity does not cause undue dyspnea or fatigue, chest pain or near syncope), Class II (slight limitation of physical activity, ordinary physical activity cause undue dyspnea or fatigue, chest pain or near syncope), Class III (marked limitation of physical activity, less than ordinary activity cause undue dyspnea or fatigue, chest pain or near syncope) and Class IV (cannot perform a physical activity without any symptoms, dyspnea and/or fatigue may even be present at rest). Change from baseline in WHO functional class was classified into "Improved", "No change" and "Worsened". Improvement =reduction in functional class; worsened =increase in functional class; and no change = no change in functional class.
Time Frame: Baseline, Week 26
Population: Safety analysis set included all participants who received at least 1 dose of study intervention. Here, "N" (Overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 8
Participants
  Baseline: Class I | 0
  Baseline: Class II | 4
  Baseline: Class III | 4
  Baseline: Class IV | 0
  Week 26: Improved | 3
  Week 26: Unchanged | 5
  Week 26: Worsened | 0

8. Secondary Outcome: Change From Baseline to Week 26 in N-terminal-Pro-Hormone Brain Natriuretic Peptide (NT-proBNP)
Description: NT pro-BNP is a cardiac biomarker that is released in the blood in response to changes in the pressure inside of the heart. Levels go up when heart failure develops or gets worse, and levels go down when heart failure is stable or improves. This biomarker helps to measure the changes in the severity of heart failure over time in response to therapy.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: nanograms/liter (ng/L)
Arm/Group | Selexipag
Number analyzed (Participants) | 6
nanograms/liter (ng/L)
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | -202.376
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 142.9233
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | -261.4904
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 78.6501
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | -215.8226
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | -762.5677

9. Secondary Outcome: Change From Baseline to Week 26 in 6-Minute Walk Distance (6MWD)
Description: 6MWD was the distance that a participant could walk in 6 minutes. Participants were asked to perform the test at a pace that was comfortable to them, with as many breaks as they needed.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Meter
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Meter
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | -72
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 275
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 14
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 17
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 16

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product. Any AE occurring at or after the initial administration of study intervention up to 3 days after last dose of study intervention was considered as treatment-emergent.
Time Frame: Day 1 up to 3 days after last dose of study drug (up to 52 weeks and 3 days that is 367 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 9
Participants
  AEs | 9
  SAEs | 1

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Premature Discontinuation of Study Drug
Description: Number of participants with AEs leading to premature discontinuation of study drug were reported. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Day 1 up to last dose of study drug (up to Week 52)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 9
Participants | 0

12. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: Number of participants with AESI were reported. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AESI were anaemia, bleeding events, gastrointestinal disturbances denoting intestinal intussusception (manifested as ileus or obstruction), hyperthyroidism, hypotension, light-dependent non-melanoma skin malignancies, major adverse cardiovascular events (MACE), medication errors, ophthalmological effects associated to retinal vascular system, pregnancy, pulmonary venoocclusive disease associated with pulmonary oedema, renal function impairment / acute renal failure.
Time Frame: Day 1 up to 3 days after last dose of study drug (up to 52 weeks and 3 days that is 367 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 9
Participants | 3

13. Secondary Outcome: Number of Participants With Treatment-Emergent Marked Laboratory Abnormalities
Description: Number of participants with treatment-emergent marked laboratory abnormalities in alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, creatinine, sodium, potassium, hemoglobin, hematocrit; EVF; PCV (male), hematocrit; EVF; PCV (female), platelets (assuming no platelet cluster), leukocytes; white blood cells, Neutrophils (Abs), Eosinophils (Abs), lymphocytes (Abs) were reported. Abnormalities that occurred after study treatment start and up to 3 days after study treatment discontinuation, that were not present at baseline, were treatment-emergent. Treatment-emergent marked laboratory abnormalities were determined at the investigator's discretion.
Time Frame: Day 1 up to 3 days after last dose of study drug (up to 52 weeks and 3 days that is 367 days)
Population: Safety analysis set included all participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Selexipag
Number analyzed (Participants) | 9
Participants | 3

14. Secondary Outcome: Change From Baseline to Week 26 in Number of Non-invasive Low-risk Criteria Among the 8 Variables
Description: The risk score is derived for each participant considering the following non-invasive low-risk criteria among the 8 variables: absence of clinical signs of right heart failure, absence of symptoms progression, absence of syncope, WHO FC I-II, 6MWD greater than (>) 440 meter, NT-proBNP less than (<) 300 ng/L, Right atrial (RA) area <18 centimeter square (cm^2) as determined by echocardiography (Echo), absence of pericardial effusion, as determined by Echo. Number of low-risk criteria at baseline and Week 26 constitutes risk score and were derived for each participant by adding '1' for each of above criteria met. Number of low-risk criteria among the 8 variables for each participant can vary from 0 (worse participants) to 8 (healthier participants). Higher score indicated healthier participants.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Score on a scale
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Score on a scale
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 1
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 3
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 1
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 1
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 1

15. Secondary Outcome: Change From Baseline to Week 26 in Number of Non-invasive Low-risk Criteria Among the 3 Variables
Description: The risk score is derived for each participant considering the following non-invasive low-risk criteria among the 3 variables: WHO FC I-II, 6MWD >440 m, NT-proBNP < 300 ng/L. Number of low-risk criteria at baseline and Week 26 constitutes risk score and were derived for each participant by adding '1' for each of above criteria met. Number of low-risk criteria among the 3 variables for each participant can vary from 0 (worse participants) to 3 (healthier participants). Higher score indicated healthier participants.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Number; unit: Score on a scale
Arm/Group | Selexipag
Number analyzed (Participants) | 6
Score on a scale
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 0
  Participant 3: number analyzed (Participants) | 1
  Participant 3 | 2
  Participant 4: number analyzed (Participants) | 1
  Participant 4 | 1
  Participant 5: number analyzed (Participants) | 1
  Participant 5 | 1
  Participant 6: number analyzed (Participants) | 1
  Participant 6 | 1

ADVERSE EVENTS:
Time Frame: All Cause Mortality: Day 1 up to 30 days after last dose of drug (up to Week 56), SAEs and non-SAEs: Day 1 up to 3 days after last dose of study drug (up to 52 weeks and 3 days that is 367 days)
Description: Safety analysis set included all participants who received at least 1 dose of study intervention.
Arm/Group | Selexipag
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=9)
Cardiac Failure (Cardiac disorders) | 1 (1)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selexipag (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Xerophthalmia (Eye disorders) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (8)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 7 (8)
Vomiting (Gastrointestinal disorders) | 2 (3)
Chest Pain (General disorders) | 2 (2)
Face Oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Oedema Peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Covid-19 (Infections and infestations) | 3 (3)
Fungal Skin Infection (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Body Temperature Increased (Investigations) | 1 (1)
Vitamin D Decreased (Investigations) | 1 (1)
Weight Decreased (Investigations) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness Exertional (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (7)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (2)
Renal Pain (Renal and urinary disorders) | 1 (1)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Flushing (Vascular disorders) | 2 (2)
Hot Flush (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT04435782/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT04435782/SAP_001.pdf